CLINICAL TRIAL: NCT06155955
Title: Comparison of Outcomes Between Low Dose Emicizumab and Extended Half-life Factor VIII With Pharmacokinetic-guided Prophylaxis in Clinically Severe Hemophilia A
Brief Title: Comparison of Outcomes Between Low Dose Emicizumab and Factor VIII in Clinically Severe Hemophilia A
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Nuchanun Kessakorn, MD, MD, Chulalongkorn University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KingChulalongkorn
Record Dates: First submitted 2023-11-11; First posted 2023-12-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Severe Hemophilia A Without Inhibitor; Joint Bleed
Keywords: emicizumab; hemophilia A
MeSH Terms: conditions — Hemarthrosis; Hemophilia A | interventions — emicizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low dose emicizumab (Experimental): 2 mg per kilograms per dose in first month, loading every 2 weeks then every 4 weeks
  Interventions: Drug: "Emicizumab", "HEMLIBRA®"
- low dose factor VIII prophylaxis (No Intervention): factor VIII prophylaxis

INTERVENTIONS:
Drug: "Emicizumab", "HEMLIBRA®" — low dose
  Other Names: emicizumab-kxwh
  Arms: low dose emicizumab

SUMMARY:
* To outcome between low dose Emicizumab and low dose prophylaxis with FVIII concentration
* To study pharmacokinetic, side effect of low dose Emicizumab

DETAILED DESCRIPTION:
* To compare outcome between low dose Emicizumab and low dose prophylaxis with FVIII concentration using ABR, AJBR and HJHS, HaemoQoL
* To study pharmacokinetic, side effect and effectiveness of low dose Emicizumab

ELIGIBILITY:
Inclusion Criteria:

* Severe or moderate Hemophilia A with baseline FVIII:C of <3 IU/dl or severe bleeding phenotype
* Receiving low dose FVIII prophylaxis for at least 6 months

Exclusion Criteria:

* Detectable FVIII inhibitor at screening
* Detectable FVIII inhibitor at screening Having other underlying diseases: Juvenile rheumatoid arthritis, metabolic bone diseases, or other conditions mimicking or causing joint diseases

Ages: 3 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-06-22 (Actual); Primary Completion 2024-03-21 (Estimated); Study Completion 2024-06-21 (Estimated)

PRIMARY OUTCOMES:
spontaneous and traumatic bleeding rate | 6 months after start low dose emicizumab as secondary prophylaxis treatment
  Using "Annualized bleeding rate" (ABR)
treated spontaneous bleeds, treated joint bleeds | 6 months after start low dose emicizumab as secondary prophylaxis treatment
  Using "Annualized joint bleeding rate" (AJBR)
The function of the knee, elbow, and ankle joints | 6 months after start low dose emicizumab as secondary prophylaxis treatment
  Using "Hemophilia Joint Health Score" (HJHS)

CONTACTS AND LOCATIONS:
Overall Officials: NUCHANUN KESSAKORN, Principal Investigator — King Chulalongkorn Memorial Hospital
Locations (1):
- King Chulalongkorn Memorial hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kessakorn N, Gosriwatana I, Sasipong N, Srichumpuang C, Moonla C, Sosothikul D. Low-Dose Emicizumab Versus Low-/Intermediate-Dose Factor VIII Secondary Prophylaxis for Noninhibitor Haemophilia A Patients With Severe Bleeding Phenotype. Haemophilia. 2025 Jan;31(1):122-131. doi: 10.1111/hae.15146. Epub 2024 Dec 31. PMID 39737816

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-24): https://cdn.clinicaltrials.gov/large-docs/55/NCT06155955/Prot_SAP_000.pdf